CLINICAL TRIAL: NCT03950921
Title: Improving Risk Detection and Communication to Reduce Hospital-Acquired Conditions
Brief Title: Pilot Testing a Patient Safety Display in the Hospital Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer Meddings, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00106108
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Catheter-Related Infections; Pressure Injury
Keywords: Catheter-Related Infections; Pressure Injury; Patient Safety
MeSH Terms: conditions — Catheter-Related Infections; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Intervention-control study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Safety Display Arm (Experimental): Patient Safety Display in patient room
  Interventions: Behavioral: Patient Safety Display
- Control Arm (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Patient Safety Display — Digital display of catheter and pressure injury information in patient hospital room
  Arms: Patient Safety Display Arm

SUMMARY:
This is a feasibility pilot study to introduce and evaluate an intervention designed to increase clinician awareness of their patients' urinary catheters, vascular catheters, and pressure injuries. This intervention, the "Patient Safety Display" will be evaluated in one hospital unit.

DETAILED DESCRIPTION:
This project will introduce and evaluate an intervention designed to increase clinician awareness of their patients' urinary catheters, vascular catheters, and pressure injuries. A "Patient Safety Display" will be implemented in half of the patient rooms in one hospital unit. The Patient Safety Display will display catheter and pressure injury data pulled real-time from the electronic medical record onto a tablet mounted at the patient bedside.

This is an intervention-control design study that will be conducted with patients and clinicians at Michigan Medicine. The proposed intervention, the Patient Safety Display, will provide clinicians with key catheter and skin information at the bedside when pertinent clinical decisions are being made.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in specific hospital unit of interest or providers caring for patient in that unit

Exclusion Criteria:

* Patients not in unit of interest and providers not caring for patients on that unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Urinary catheter awareness | 4 months
  Proportion of physicians and advanced practice providers aware of their patients' indwelling urinary catheters; measured via survey
Central venous catheter awareness | 4 months
  Proportion of physicians and advanced practice providers aware of their patients' central venous catheters; measured via survey
Pressure injury awareness | 4 months
  Proportion of physicians and advanced practice providers aware of their patients' pressure injuries; measured via survey

SECONDARY OUTCOMES:
Urinary catheter usage | 4 months
  Urinary catheter usage rates, as documented in the electronic medical record
CAUTI | 4 months
  Catheter-associated urinary tract infections (CAUTI) rates, as collected for routine National Healthcare Safety Network (NHSN) reporting
Central venous catheter usage | 4 months
  Central venous catheter usage rates, as documented in the electronic medical record
CLABSI | 4 months
  Central-line associated urinary tract infections (CLABSI) rates, as collected for routine NHSN reporting
Pressure injuries | 4 months
  Pressure injury incidence, as documented in the electronic medical record
Pressure injury care | 4 months
  Rates of pressure injury care practices (i.e., wound team consults, specialty bed orders, use of repositioning devices) as reported in the electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Meddings, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University Hospital, Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No